CLINICAL TRIAL: NCT01387971
Title: Using Impression Cytology to Observe the Cytological Changes of Ocular Surface Cells in Various Ocular Surface Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: We-Li Chen , MD, Natinal Taiwan University Hospital
Other Study IDs: 200910001R
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-04

CONDITIONS: Pterygium; Dry Eye; Tumor
Keywords: impression cytology; ocular surface disorders; ocular surface cells' variation; Limbal insufficiency
MeSH Terms: conditions — Pterygium; Dry Eye Syndromes; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ocular surface disorders: various ocular surface disorders

SUMMARY:
Currently, due to the advantage of noninvasive, localized, rapid, painless and easily repeatable of impression specimens, the technique is an ideal method of investigating ocular surface disorders when the diagnosis is not clinically obvious or detecting the post-operative change without tissue damage. Using impression cytology for primary diagnosis and follow-up of ocular surface squamous neoplasia, including after therapy with topical mitomycin C has been well-studied. [29]. In addition to the applications described above, pterygium is another disease of interest. Pterygium, a common disease of ocular surface, has high recurrence rate after surgical excision. [30-33] However, the exact etiology and mechanism for recurrence is unknown. A transformation of the phenotypic characteristics of the conjunctival fibroblasts may play an important role. Due to the concern of improvement in treatment, it is important to explore the change of cytomorphology after pterygium operation, to identify the risk factors of developing recurrence, and, furthermore, to clarify the etiology and mechanism. Some ophthalmologists may think this procedure too time-consuming to be a routine examination in outpatient clinics. [34] However, National Taiwan University Hospital (NTUH), as one of the largest tertiary medical centers in Taiwan, is now in charge of a big part of difficult cases of ocular surface. With the need of further precise diagnosis and delicate clinical skills, the investigators are competent for this meaningful program.

DETAILED DESCRIPTION:
Impression cytology is a simple, noninvasive technique that has been widely used to aid in the diagnosis of several disorders of the ocular surface. The first use of impression cytology specimens for diagnosis of ocular surface squamous neoplasia was reported in France in 1954 by Larmande and Timsit. [1] In the English language literature, Egbert et al [2] in 1977 documented the use of cellulose acetate filters to detect goblet cell density in patients with the dry eye syndrome. Traditionally, the cytology specimens were obtained by pressing cellulose acetate (Millipore) filters onto the surface of the globe, then air-dried and stained with PAS. [2] The procedure is usually painless even without anesthesia. The filters remove 1 to 3 superficial cell layers of conjunctiva and cornea.

Since its first applications in ocular surface squamous neoplasia and dry eye syndrome, [1,2] the use of impression cytology has expanded to include the staging of conjunctival squamous metaplasia, [3,4] diagnosis of ocular surface squamous neoplasia, [5-11] and follow-up of ocular surface squamous neoplasia after topical mitomycin-C, [10] limbal stem-cell deficiency, [12,13] specific viral infections, [14-16] vitamin A deficiency, [17,18] epithelial cell storage disorders, [19] allergic disorders, [19] conjunctival melanosis and malignant melanoma, [20] and psoriasis [21]. The technique has the additional advantage of preserving limbal stem cells, which occur in the basal layer of the limbal epithelium and are responsible for renewal of the corneal epithelium throughout life. Since ocular surface squamous neoplasia preferentially involves the limbus, limbal stem cells are potentially reduced in number with each surgical biopsy. The progressive loss of limbal stem cells results in limbal stem-cell deficiency, conjunctivalization of the cornea with corneal opacity. Thus, impression cytology offers a safer alternative to diagnosis than repeated biopsies.

With impression cytology, the morphology of the corneal and conjunctival epithelial cells, their staining behavior, and nuclear/cytoplasmic ratio could be observed in detail. Other important characteristics such as goblet cell density, the degree of keratinization of the epithelial cells, the quality of the cell-to-cell cohesion, and the condensation of the nuclear chromatin could also be detected through proper specimens. [3, 22-26] Furthermore, with the improvement of immunocytochemical staining and confocal microscopy, specimens of impression cytology can be further analyzed for complicated ocular disorder such as cytokeratins 3 and 19 are useful in classification of limbal stem cell deficiency [27] and mucin secretion of goblet cells can be evaluated by confocal microscopy [28].

ELIGIBILITY:
Inclusion Criteria:

* various ocular surface disorders

Exclusion Criteria:

1. cognitive function disorder
2. extremely ocular surface discomfort

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: various ocular surface disorders
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, PhD, Principal Investigator — National Taiwan University Hospital, department of Ophthalmology
Locations (1):
- National Taiwan University Hospital, department of Ophthalmology, Taipei, Taiwan, Taiwan